CLINICAL TRIAL: NCT07193225
Title: Non-invasive Mapping of Coronary Arteries and the Cerebral Vascular Network Using 3D Ultrasound Localization Microscopy in Patients With Atherosclerosis Prior to Carotid Endarterectomy Surgery - Microflow3D
Brief Title: Microflow3D - Non-invasive Mapping of Coronary Arteries and the Cerebral Vascular Network Using 3D Ultrasound Localization Microscopy in Patients With Atherosclerosis Prior to Carotid Endarterectomy Surgery
Acronym: Microflow3D
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-01
Record Dates: First submitted 2025-09-18; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Carotid Atherosclerosis
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Intervention Model Description: Exploratory investigation, first in human, one center, open study,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ultrasound localization microscopy (Experimental): The research protocol is integrated into the patient's routine preoperative visit. During this visit, the patient undergoes echocardiography and Doppler ultrasound of the supra-aortic trunks combined with transcranial Doppler. The use of microbubbles (SonoVue®) as a contrast agent is common in cases of poor visualization. We propose to add dedicated ultrasound localization microscopy sequences coupled with SonoVue® injection during this examination in order to image the circle of Willis and the coronary arteries.
  Interventions: Device: Ultrasound localization microscopy, circle of Willis; Device: Ultrasound localization microscopy, coronary arteries

INTERVENTIONS:
Device: Ultrasound localization microscopy, circle of Willis — Ultrasound localization microscopy sequences coupled with SonoVue® injection of the circle of Willis before carotid endarterectomy
Device: Ultrasound localization microscopy, coronary arteries — ultrasound localization microscopy sequences coupled with SonoVue® injection of coronary arteries before carotid endarterectomy

SUMMARY:
There is a need to simplify the assessment of coronary and cerebral vascular networks in patients selected for carotid endarterectomy in order to prevent potential complications during and after surgery. A non-invasive, non-ionizing 3 dimension mapping of these networks would provide a remarkable benefit for patients.

DETAILED DESCRIPTION:
Carotid atherosclerosis is associated with a high risk of stroke due to embolization from vulnerable plaques located at the carotid bifurcation. When the degree of stenosis exceeds 60%, carotid endarterectomy is considered to remove the plaque. This is a complex surgical procedure, performed under general anesthesia in most cases, and consists of extracting the plaque. The patient population is typically elderly and particularly fragile, with a significant risk of cerebral infarction during the intervention. To minimize perioperative risks, patients undergo a preoperative evaluation that includes transcranial Doppler ultrasound and coronary angiography. The purpose of transcranial Doppler is to image the circle of Willis and identify patients with an incomplete circle, which would compromise adequate cerebral perfusion during carotid clamping. However, this imaging is challenging because the quality of ultrasound through the skull is often poor, and two-dimensional imaging does not always allow full visualization of the circle of Willis. A high-resolution three-dimensional imaging modality could therefore improve surgical planning. Coronary angiography or CT coronary angiography are performed to image the coronary arteries and identify patients at highest risk of myocardial infarction. A non-ionizing three-dimensional imaging modality with high coronary resolution could also benefit patients by reducing radiation exposure.

Ten years ago, the Physics for Medicine Laboratory developed a novel imaging technique called ultrasound localization microscopy (ULM). This modality combines ultrafast ultrasound imaging (acquiring more than 1000 frames per second) with the injection of microbubbles already used in clinical practice. By individually imaging and localizing these microbubbles, it becomes possible to visualize the vascular networks of the coronary arteries and the brain in animal models with unprecedented resolution and field of view. Recently, the clinical feasibility of ultrasound localization microscopy was demonstrated in two dimensions in the brain of patients with cerebral aneurysms.

Nevertheless, the two-dimensional nature of the imaging represented a limitation. To address this, we developed a new type of wider ultrasound probe capable of imaging large three-dimensional volumes. These probes have already been validated through simulations, phantom studies, and more recently in animal experiments.

In this clinical study, we therefore aim to demonstrate the feasibility of three-dimensional imaging of the microcirculation of the heart and brain in patients during the preoperative evaluation, with the goal of improving surgical planning for carotid endarterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with asymptomatic carotid stenosis, without recent stroke, and scheduled for carotid endarterectomy within the next 30 days.
* Age ≥ 18 years.
* Beneficiary of a social security system or equivalent coverage.
* Signed informed consent.
* Patients already enrolled in another biomedical research study may also participate in this study.

Exclusion Criteria:

* Contraindication to the use of the ultrasound contrast agent SonoVue®: known hypersensitivity to the active substance or to any of the following excipients: Macrogol 4000; Distearoylphosphatidylcholine; Sodium dipalmitoylphosphatidylglycerol; Palmitic acid.
* Allergy to ultrasound gel.
* Refusal or inability (linguistic or psychological) to sign the informed consent form.
* Subject to legal protection measures, such as guardianship (in accordance with Article L1122-2 of the French Public Health Code).
* Pregnant or breastfeeding women cannot participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Detecting the presence of an incomplete circle of Willis | At day 0
  Detection of all arteries of the circle of Willis using ultrasound localization microscopy, compared with cerebral Computed Tomography angiography or Magnetic Resonance Imaging, routinely performed before carotid endarterectomy.

SECONDARY OUTCOMES:
Detecting the presence of coronary stenosis | At day 0
  Detection of coronary stenosis using ultrasound localization microscopy, compared with coronary Computed Tomography angiography or coronary angiography, routinely performed before carotid endarterectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume GOUDOT, MD, Study Chair — APHP, Georges Pompidou European Hospital, France; Clément PAPADACCI, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Georges Pompidou European Hospital, Paris, France